CLINICAL TRIAL: NCT04431960
Title: Blackcurrant Modifies Gut Microbiota and Reduces the Risk of Postmenopausal Osteoporosis and Cardiovascular Disease: A Pilot Randomized Clinical Trial
Brief Title: Blackcurrants Modify Gut Microbiota and Reduce Osteoporosis and CVD Risk
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Ock Chun, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HR20-0035; 2020-67018-30852 (Other Grant/Funding Number: USDA NIFA)
Record Dates: First submitted 2020-06-06; First posted 2020-06-16 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Postmenopausal Osteoporosis; Gut Microbiota; Cardiovascular Diseases
Keywords: blackcurrant; gut microbiome; osteoporosis; menopause; bone aging; women; cardiovascular disease
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Cardiovascular Diseases; Osteoporosis

STUDY DESIGN:
Intervention Model Description: The study participants will be randomly assigned to three groups and asked to consume 1 tablet containing 392 mg blackcurrant (BC) extract per capsule (low-BC Group), 2 capsules containing 392 mg BC extract per tablet (total 784 mg/day; high-BC Group), or 1 placebo capsule (Control Group) daily with breakfast meals for 6 months.
  To avoid bone deterioration related to calcium and vitamin D deficiency, all participants will take a calcium citrate caplet daily that includes 400 mg calcium and 500 IU vitamin D (Bayer AG, Germany) beginning 2 weeks before the study and lasting for the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The extract and placebo will have the identical shape and color and will be packaged into coded containers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- low-BC Group (Active Comparator): consume: 1) one tablet containing 392 mg blackcurrant (BC) extract per capsule and 2) one calcium citrate caplet containing 400 mg calcium and 500 IU vitamin D
  Interventions: Drug: blackcurrant (BC) extract
- high-BC Group (Active Comparator): consume: 1) two capsules containing 392 mg BC extract per tablet (total 784 mg/day) and 2) one calcium citrate caplet containing 400 mg calcium and 500 IU vitamin D
  Interventions: Drug: blackcurrant (BC) extract
- Control Group (Placebo Comparator): consume: 1) one placebo capsule and 2) one calcium citrate caplet containing 400 mg calcium and 500 IU vitamin D
  Interventions: Drug: blackcurrant (BC) extract

INTERVENTIONS:
Drug: blackcurrant (BC) extract — A calcium citrate caplet (Bayer AG, Germany) will be taken by all 3 groups to avoid bone deterioration related to calcium and vitamin D deficiency
  Other Names: BPE75 (392 mg and 784 mg)

SUMMARY:
Aim to evaluate the effects of blackcurrant supplementation on changes in gut microbiome, bone mass, and CVD risk factors in adult women.

DETAILED DESCRIPTION:
Postmenopausal bone loss is a primary contributor to osteoporosis and osteoporotic fractures in adult women in menopause transition. By following women over this period, studies have documented distinct patterns of a decrease in estrogen, a natural antioxidant, simultaneously with adverse alterations in body fat distribution, lipids and lipoproteins, and measures of vascular health, which can increase a woman's risk of developing CVD. Overall goal of this project is to evaluate the effects of blackcurrant (BC) supplementation on changes in gut microbiome, bone mass, and CVD risk factors in adult women. For this purpose, the investigators will conduct a pilot randomized placebo-controlled clinical trial with BC supplementation for 6 months in peri- and early postmenopausal women aged 45-60 years.

The primary endpoint will be whole-body bone mineral density (BMD); secondary endpoints will be gut microbiota composition. To delineate the underlying mechanisms of the action, changes in biomarkers for bone metabolism, bone-related immune and endocrine systemic biomarkers, and CVD risk factors by BC supplementation will be measured in plasma and peripheral blood derived mononuclear cells.

The specific objectives of the study are to investigate the effects of BC extract on: 1) bone mass and bone remodeling markers; 2) changes in the gut microbiota abundance and composition, immune and endocrine biomarkers, and CVD risk factors and their relationships with changes in bone mass.

The proposed study will provide novel insight into whether and how BC consumption reduces the risk of postmenopausal bone loss and CVD in adult women and will improve understanding of the clinical roles of gut microbiome in postmenopausal bone loss. Findings from this study will help increase awareness of the bone and heart health promoting effect of BC and motivate increased production of BC and other berry products in response to the increasing consumer demand.

ELIGIBILITY:
Inclusion Criteria:

* perimenopausal or early postmenopausal women aged 45-60 years old
* not on HRT for at least one year before the initiation of the study
* maintaining normal exercise level (<7 h/wk) and willing to avoid exercise 24-h prior to blood and stool sampling and 12-h prior to bone measurements
* willing to ingest a dietary BC supplement or placebo (up to 900 mg/day, two 450 mg capsules) as well as 400 mg calcium and 500 IU vitamin D daily
* willing to avoid other dietary supplements for the duration of the study
* willing to avoid intake of foods extremely rich in anthocyanins and fermented dairy products containing viable Bifidobacteria or Lactobacilli
* willing to have 3 blood draws, 2 stool collections, and 2 bone scans
* willing to take urine pregnancy test if they are perimenopausal.

Exclusion Criteria:

* those with metabolic bone disease, renal disease, cancer, cardiovascular disease, diabetes mellitus, respiratory disease, gastrointestinal disease, liver disease or other chronic diseases
* those with hypertension or on drugs that lower blood pressure
* those with planned surgery during the study period or within 2 weeks of ending the intervention
* taking medications that alter bleeding (such as antiplatelets or anticoagulants) or those with a bleeding disorder
* taking a phenothiazine drug (most commonly used for nausea or mental health conditions)
* having a sensitivity or allergy to any of ingredients for the placebo (rice powder) and calcium/D supplement (calcium citrate, polyethylene glycol, croscarmellose sodium, hydroxypropyl methylcellulose, magnesium stearate, oligofructose enriched inulin, propylene glycol dicaprylate/dicaprate, talc, titanium dioxide, vitamin D3)
* heavy smokers (>20 cigarettes/day)
* perimenopausal women with any chance or plan of pregnancy
* taking prescription medications known to alter bone and Ca metabolism such as calcitonin, bisphosphonates, raloxifene within 3 months before the start of the study
* taking anabolic agents such as parathyroid hormone, growth hormone, or steroids within 3 months before the start of the study
* planning any procedure that includes iodine, barium or nuclear medicine isotopes in next 7 months
* alcohol consumption exceeding 2 drinks/day (approximately 14 g ethanol per drink) or a total of 12/week
* UConn students and/or employees who any key personnel teach or who report to any key personnel
* study key personnel, spouses of key personnel, or dependents/relatives of any key personnel.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — perimenopausal or early postmenopausal women
Enrollment: 51 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ock K Chun, PhD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut Department of Nutritional Sciences and Kinesiology Human Performance Laboratory, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Once research proceedings and manuscripts are published we will make our results available both to the community of scientists interested in postmenopausal osteoporosis and to those studying the biology of inflammation-induced bone resorption to avoid unintentional duplication of research.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Unlimited time after papers are published.
Access Criteria: Our plan of sharing of data generated by this project includes the following:
  1. Presentations at national scientific meetings. From the projects, it is expected that approximately two presentations at national meetings would be appropriate.
  2. Publication in peer-reviewed journals. It is our explicit intention that the study findings and key data will be placed in a readily accessible public database. All efforts will be made to rapidly release data through publication of results as quickly as possible following our analysis of the experiment data. Data used in publications will be released in a timely manner.

REFERENCES:
- [Derived] Nosal BM, Thornton SN, Darooghegi Mofrad M, Sakaki JR, Mahoney KJ, Macdonald Z, Daddi L, Tran TDB, Weinstock G, Zhou Y, Lee EC, Chun OK. Blackcurrants shape gut microbiota profile and reduce risk of postmenopausal osteoporosis via the gut-bone axis: Evidence from a pilot randomized controlled trial. J Nutr Biochem. 2024 Nov;133:109701. doi: 10.1016/j.jnutbio.2024.109701. Epub 2024 Jul 15. PMID 39019119

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-BC Group | High-BC Group | Control Group
Started | 17 | 16 | 18
Completed | 16 | 11 | 13
Not Completed | 1 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-BC Group | High-BC Group | Control Group | Total
Number analyzed (Participants) | 16 | 11 | 13 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 11 | 13 | 40
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (4.5) | 50.9 (4.2) | 54.4 (3.8) | 53.1 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 13 | 40
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ethnicity: Caucasian | 13 | 11 | 13 | 37
  Race/ethnicity: Hispanic | 1 | 0 | 0 | 1
  Race/ethnicity: Asian-American/Pacific Islander | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 16 | 11 | 13 | 40

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density (BMD)
Description: Changes in BMD of whole-body measured via dual energy x-ray absorptiometry
Time Frame: From baseline to 6 months
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Low-BC Group | High-BC Group | Control Group
Number analyzed (Participants) | 16 | 11 | 13
g/cm^2
  Baseline | 1.14 (0.13) | 1.15 (0.08) | 1.17 (0.13)
  6 month | 1.14 (0.12) | 1.17 (0.08) | 1.16 (0.13)

2. Secondary Outcome: Serum Marker of Bone Formation
Description: Changes to serum concentrations of P1NP
Time Frame: From baseline to 6 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Low-BC Group | High-BC Group | Control Group
Number analyzed (Participants) | 16 | 11 | 13
ng/mL
  Baseline | 26.55 (10.43) | 21.21 (10.09) | 32.53 (20.93)
  6 months | 25.99 (10.27) | 41.79 (39.47) | 26.36 (17.71)

3. Secondary Outcome: Plasma Regulator of Bone Metabolism
Description: Changes to plasma concentrations RANKL
Time Frame: From baseline to 6 months
Population: Analysis was performed on 35 participants for RANKL due to missing values.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low-BC Group | High-BC Group | Control Group
Number analyzed (Participants) | 15 | 10 | 10
pg/mL
  Baseline | 211.12 (89.94) | 133.99 (111.89) | 256.81 (110.39)
  6 months | 210.15 (90.43) | 102.09 (112.51) | 284.47 (111.00)

4. Secondary Outcome: Changes in Plasma Inflammatory Cytokine
Description: Changes to plasma concentrations of IL-1B
Time Frame: From baseline to 6 months
Population: Analysis was performed on 36 participants for IL-1β due to missing values.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Low-BC Group | High-BC Group | Control Group
Number analyzed (Participants) | 15 | 9 | 12
pg/mL
  Baseline | 16.73 (1.85) | 15.36 (2.44) | 17.95 (2.09)
  6 months | 16.66 (1.85) | 15.06 (2.44) | 18.34 (2.09)

5. Other Pre Specified Outcome: Changes in Gut Microbial Composition
Description: This was measured using alpha diversity by species richness and Shannon diversity and beta diversity by principal component analysis. Structural comparisons were done comparing relative abundance between groups at the genus and phylum levels
Time Frame: from baseline to 6 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Serum Inflammation Biomarker
Description: changes in serum inflammation biomarker (hs-CRP)
Time Frame: from baseline to 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Fasting Blood Lipids
Description: Changes in plasma CVD risk factors (total cholesterol [TC], high density lipoprotein [HDL] and triglycerides [TG])
Time Frame: from baseline to 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Low-BC Group | High-BC Group | Control Group
Number analyzed (Participants) | 14 | 11 | 13
mg/dL
  TC (baseline) | 179.7 (9.5) | 194.0 (10.8) | 178.1 (9.9)
  TC (3 months) | 177.5 (9.1) | 196.7 (10.2) | 180.5 (9.4)
  TC (6 months) | 167.6 (9.7) | 194.2 (11.0) | 184.0 (10.1)
  HDL (baseline) | 62.0 (4.2) | 70.8 (4.7) | 71.5 (4.3)
  HDL (3 months) | 62.9 (4.7) | 71.6 (5.3) | 72.3 (4.8)
  HDL (6 months) | 59.9 (4.5) | 73.5 (5.0) | 72.8 (4.6)
  TG (baseline) | 112.8 (10.8) | 78.1 (12.2) | 68.4 (11.2)
  TG (3 months) | 106.5 (9.6) | 87.4 (10.9) | 75.5 (10.0)
  TG (6 months) | 112.3 (8.8) | 68.9 (10.0) | 74.2 (9.2)

8. Other Pre Specified Outcome: Blood Pressure (SBP/DBP), BMI, WC, Body Composition
Description: changes in blood pressure (SBP/DBP), BMI, WC, body composition
Time Frame: from baseline to 6 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Concentrations of Plasma Immune Markers
Description: changes in plasma concentrations of immune biomarkers (IL-1β, IL-6, TNFα, Th17 and Treg)
Time Frame: from baseline to 6 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Concentrations of Plasma IGF-1 and cGP
Description: changes in plasma concentrations of endocrine biomarkers
Time Frame: from baseline to 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6.5 months total. All participants took a calcium citrate caplet daily that includes 400 mg calcium and 500 IU vitamin D beginning 2 weeks before the study and lasting for the duration of the study. After the 2-week equilibration period, study participants were randomly assigned to three groups and asked to consume the provided intervention drug daily for 6 months.
Description: During the entire study period and at each study visit, participants were asked by research staff to report if they experience any adverse events from the intervention.
Arm/Group | Low-BC Group | High-BC Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/16 | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT04431960/Prot_SAP_000.pdf